CLINICAL TRIAL: NCT04797793
Title: A Double-blind, Randomized, Placebo Controlled Study to Compare Adapalene Gel 0.1% to Differin Gel and Both Active Treatments to a Placebo Control in the Treatment of Acne Vulgaris
Brief Title: A Study Comparing Adapalene Gel 0.1% and to Differin Gel in the Treatment of Acne Vulgaris
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ADBG-2043
Record Dates: First submitted 2021-03-12; First posted 2021-03-15 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Adapalene

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Adapalene gel 0.1% (Experimental): The study medication will be self-applied topically, on the affected areas of the face lightly, once daily at bedtime, avoiding contact with the mouth, eyes, and other mucous membranes for 84 consecutive days.
  Interventions: Drug: Adapalene Gel 0.1%
- Differin® Gel (Adapalene 0.1%, Galderma) (Active Comparator): The study medication will be self-applied topically, on the affected areas of the face lightly, once daily at bedtime, avoiding contact with the mouth, eyes, and other mucous membranes for 84 consecutive days.
  Interventions: Drug: Differin® Gel (Adapalene 0.1%, Galderma)
- Placebo Control (Placebo Comparator): The study medication will be self-applied topically, on the affected areas of the face lightly, once daily at bedtime, avoiding contact with the mouth, eyes, and other mucous membranes for 84 consecutive days.
  Interventions: Drug: Placebo Control

INTERVENTIONS:
Drug: Adapalene Gel 0.1% — The study medication will be self-applied topically on the affected areas of the face lightly, once daily at bedtime, avoiding contact with the mouth, eyes, and other mucous membranes for 84 consecutive days.
  Other Names: Test Product
  Arms: Adapalene gel 0.1%
Drug: Placebo Control — The study medication will be self-applied topically on the affected areas of the face lightly, once daily at bedtime, avoiding contact with the mouth, eyes, and other mucous membranes for 84 consecutive days.
  Other Names: Vehicle
  Arms: Placebo Control
Drug: Differin® Gel (Adapalene 0.1%, Galderma) — The study medication will be self-applied topically on the affected areas of the face lightly, once daily at bedtime, avoiding contact with the mouth, eyes, and other mucous membranes for 84 consecutive days.
  Other Names: Reference Product
  Arms: Differin® Gel (Adapalene 0.1%, Galderma)

SUMMARY:
To demonstrate therapeutic equivalence and safety of adapalene gel 0.1% (Taro Pharmaceuticals U.S.A., Inc.) and Differin® Gel (Adapalene Gel 0.1%, Galderma) in the treatment of acne vulgaris.

DETAILED DESCRIPTION:
A multi-center, double-blind, randomized, placebo controlled, parallel-group study, Adapalene Gel 0.1% (Taro Pharmaceuticals U.S.A, Inc.) and to Differin® Gel (Adapalene 0.1%, Galderma) and both active treatments to a placebo control in the treatment of acne vulgaris

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non pregnant female aged ≥ 12 and ≤ 40 years with a clinical diagnosis of acne vulgaris.
* Subjects who are 18 years of age or older (up to the age of 40) must have provided IRB approved written informed consent. Subjects ages 12 to 17 years of age inclusive must have provided IRB approved written assent;
* Subjects must have a definite clinical diagnosis of acne vulgaris of severity grade 2, 3, or 4 as per the Investigator's Global Assessment (IGA)

Exclusion Criteria:

* Female Subjects who are pregnant, nursing or planning to become pregnant during study participation
* Subjects with a history of hypersensitivity or allergy to tretinoin, retinoids, or any of the study medication ingredients.
* Subjects with the presence of any skin condition that would interfere with the diagnosis or assessment of acne vulgaris (e.g., on the face: rosacea, dermatitis, psoriasis, squamous cell carcinoma, eczema, acneiform eruptions caused by medications, steroid acne, steroid folliculitis, or bacterial folliculitis).

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 978 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2021-01-08 (Actual); Study Completion 2021-01-08 (Actual)

PRIMARY OUTCOMES:
The percentage change in the inflammatory and non-inflammatory lesion counts | Baseline to Week 12
  Demonstration of Therapeutic Equivalence

CONTACTS AND LOCATIONS:
Overall Officials: Zaidoon A. Al-Zubaidy, Study Director — Catawba Research
Locations (1):
- Catawba Research, LLC, Charlotte, North Carolina, United States